CLINICAL TRIAL: NCT00394030
Title: An Open-Label, Randomized, Multi-Site Study to Assess the Pharmacokinetics of Single Subcutaneous Injections of 16mg and 64mg of GSK716155 Administered at Three Different Injection Sites in Adult Male and Female Subjects With Type 2 Diabetes and of Single Subcutaneous Injections of 16mg and 64mg of GSK716155 Administered in the Abdomen of Healthy, Normal Volunteers
Brief Title: Injection Site Study In Patients With Type 2 Diabetes Mellitus (T2DM) And Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP107724
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK716155 pharmacodynamics pharmacokinetics injection site
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (8):
- Group A (Experimental): In Group A healthy subjects will be randomized to receive 16 milligram (mg) of GSK716155 to abdomen.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group B (Experimental): In Group B healthy subjects will be randomized to receive 64 mg of GSK716155 to abdomen.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group C (Experimental): In Group C Type II diabetes subjects will be randomized to receive 16 mg of GSK716155 to abdomen.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group D (Experimental): In Group D Type II diabetes subjects will be randomized to receive 16 mg of GSK716155 to arm.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group E (Experimental): In Group E Type II diabetes subjects will be randomized to receive 16 mg of GSK716155 to leg.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group F (Experimental): In Group F Type II diabetes subjects will be randomized to receive 64 mg of GSK716155 to abdomen.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group G (Experimental): In Group G Type II diabetes subjects will be randomized to receive 64 mg of GSK716155 to arm.
  Interventions: Drug: GSK716155 subcutaneous injections
- Group H (Experimental): In Group H Type II diabetes subjects will be randomized to receive 64 mg of GSK716155 to leg.
  Interventions: Drug: GSK716155 subcutaneous injections

INTERVENTIONS:
Drug: GSK716155 subcutaneous injections — GSK716155 will be available as lyophilize uniform cake in 10 milliliter (mL) clear glass vials with 20 millimeter (mm) closure. Subjects will administer dose of either 16mg or 64mg of GSK716155 via subcutaneous injection(s). For dose of 16 mg 1 injection of 0.62 mL will be administered and for dose of 64 mg 3 injections of 0.82 mL each will be administered.

SUMMARY:
This study is an open-label study in healthy volunteers and in patients with Type 2 Diabetes Mellitus to assess safety and tolerability parameters, the levels of GSK716155 in the bloodstream after a single dose given at different injection sites, and the impact this medication has on various substances in the blood. Assessments include ECGs, vital signs, repeat blood sampling and monitoring of any side effects.

DETAILED DESCRIPTION:
An Open-Label, Randomized, Multi-Site Study to Assess the Pharmacokinetics of Single Subcutaneous Injections of 16mg and 64mg of GSK716155 Administered at Three Different Injection Sites in Adult Male and Female Subjects with Type 2 Diabetes and of Single Subcutaneous Injections of 16mg and 64mg of GSK716155 Administered in the Abdomen of Healthy, Normal Volunteers

ELIGIBILITY:
Inclusion criteria:

* They can be healthy volunteers or subjects with type 2 diabetes mellitus that has been diagnosed for at least three months. T2DM subjects must be taking either (1) no medication for their diabetes or (2) taking metformin or (3) taking a TZD (thiazolidinedione).
* Subjects must have a BMI between 25 and 40 kg/m² and weigh at least 50kg.
* Women must be of non-childbearing potential.

Exclusion criteria:

* Bloodwork that meets certain criteria (for example, total cholesterol > 240 mg/dL)
* Clinically significant hepatic enzyme elevation
* HbA1c less than 6.5 or greater than 10
* Positive test result for Hepatitis B surface antigen, positive Hepatitis C or HIV
* Any major illness other than diabetes
* Previous use of insulin as treatment for diabetes
* Significant renal disease as defined by screening lab tests
* History of drug or other allergy which in the opinion of the investigator contradicts subject participation
* Smoking or use of nicotine-containing products within the previous 6 months
* History of alcohol or drug abuse
* Unwilling to abstain from alcohol prior to and during the in-patient clinic stays
* Unwilling to abstain from caffeine- or xanthine-containing products prior to and during the in-patient clinic stays
* Use of St. John's Wort during the study
* Has donated 500 nL or more blood within 56 days of dosing or plans to donate blood in the month following study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-10-16 (Actual); Primary Completion 2007-03-20 (Actual); Study Completion 2007-03-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements for different injection sites after one dose. | Pre-dose, 6, 24, 48, 96, 216, 312, 480, 672 and 984 hours

SECONDARY OUTCOMES:
Pharmacodynamic measurements at three different times after one dose. | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Morrisville, North Carolina
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Results for study GLP107724 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/GLP107724?search=study&search_terms=GLP107724#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: GLP107724 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register